CLINICAL TRIAL: NCT00685048
Title: Brief Therapies for Problem Gambling Substance Abusers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 07-108-2; R01DA021567 (NIH); R01DA021567-01 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gambling
Keywords: Gambling; Brief Therapies; Substance Abuse
MeSH Terms: conditions — Gambling; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): psychoeducation
  Interventions: Behavioral: 10 minutes of psycho-education
- 2 (Experimental): brief advice
  Interventions: Behavioral: 10 minutes of brief advice
- 3 (Experimental): Motivational Enhancement Therapy (MET)/Cognitive-Behavioral Therapy (CBT)
  Interventions: Behavioral: four 50-minute individual therapy sessions of MET & CBT

INTERVENTIONS:
Behavioral: 10 minutes of psycho-education — Patients review with study therapist a brochure about types of gambling people engage in and relationships between gambling, drug use, moods, and legal problems.
  Arms: 1
Behavioral: 10 minutes of brief advice — Patients will review with study therapist a brochure and advice about problem gambling. It will also contain methods for reducing gambling.
  Arms: 2
Behavioral: four 50-minute individual therapy sessions of MET & CBT — MET & CBT
  Arms: 3

SUMMARY:
This project evaluates the efficacy of brief interventions for individuals seeking treatment for substance use disorders who also have gambling problems. In total, 220 problem gambling substance abusers will be randomized to one of three conditions: (a) a control condition consisting of 10 minutes of psychoeducation about gambling, (b) 10 minutes of brief advice about problem gambling and how to reduce it, or (c) four session of motivational and cognitive-behavioral therapy. Gambling, substance use and psychosocial problems will be assessed using standardized instruments at pre-treatment, month 2, 5, 8, 12, 16, 20 and 24-month follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* current (past-year) DSM-IV criteria for alcohol, cocaine, opioid or marijuana abuse or dependence
* score >3 on the past-two month SOGS
* report an average of >2 gambling days per month for the past 2 months; (e) spent an average of >$50/month on gambling in the past 2 months
* English speaking
* sign informed consent.

Exclusion Criteria:

* have uncontrolled major psychiatric disorders other than substance use that require inpatient hospitalization (e.g., active bipolar disorder, psychosis, suicidality)
* desire specific gambling treatment or are currently receiving treatment for gambling
* have severe cognitive impairment
* read below 5th grade level
* plan to relocate >100 miles or are likely to be incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
dollars and days gambled per month | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States